CLINICAL TRIAL: NCT06448793
Title: Patient and Physician Preferences for Potentially Resectable, Non-metastatic Non-small Cell Lung Cancer Treatments
Brief Title: Patient and Physician Preference Study in Resectable, Non-small Cell Lung Cancer Treatments
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1384
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a diagnosis of resectable non-small cell lung cancer (NSCLC)
  Interventions: Drug: Approved Non-small Cell Lung Cancer (NSCLC) therapies
- Physicians currently treating resectable non-small cell lung cancer (NSCLC) patients
  Interventions: Drug: Approved Non-small Cell Lung Cancer (NSCLC) therapies

INTERVENTIONS:
Drug: Approved Non-small Cell Lung Cancer (NSCLC) therapies — As prescribed by treating physician

SUMMARY:
The purpose of this study is to investigate the perspectives and preferences of patients and healthcare professionals (medical oncologists, pneumologists, thoracic surgeons) regarding treatment options in the resectable non-small cell lung cancer (NSCLC) setting

ELIGIBILITY:
Inclusion Criteria:

Patients

* Aged ≥18 years at the time of enrollment in the study
* Resident of the US, Germany, or Japan
* Able to read, speak, and understand English, German or Japanese
* Diagnosed with resectable phase II to IIIB non-small cell lung cancer (NSCLC)

Physicians

* Resident of the US, Germany, or Japan
* Lung cancer-treating physician specialized in one of the following medical areas: oncology, pneumonology, thoracic surgery, or radiology
* Treated at least three new patients with resectable NSCLC in the past year

Exclusion Criteria:

Patients

* Appears to have sensory and/or cognitive impairment(s) that could interfere with their ability to provide online and/or verbal consent, or complete any other interview activities (based on screener judgment)
* Being diagnosed with another malignancy alongside NSCLC
* Not willing to be audio-recorded during the interview

Physicians

* Appears to have sensory and/or cognitive impairment(s) that could interfere with their ability to provide online and/or verbal consent, or complete any other interview activities (based on screener judgment)
* Not willing to be audio-recorded during the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults participants with a diagnosis of resectable NSCLC and physicians treating patients with resectable NSCLC residing in US, Germany or Japan.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Responses to qualitative interview questions | Day 1
  Interview questions designed to gather insights into diagnosis, symptoms, current treatments, perspectives on treatment features and test for mock preferences tasks. The interview will take 15 minutes to complete.
Patient sociodemographic | Day 1
Patient clinical characteristics | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Evidera, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts